CLINICAL TRIAL: NCT07173153
Title: Phase I/II Intrathecal Gene Delivery Clinical Trial of scAAV9.P546.SLC6A1 for SLC6A1 Neurodevelopmental Disorder
Brief Title: Gene Therapy for SLC6A1 Neurodevelopmental Disorder
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Emily de los Reyes (Other)
Responsible Party: Sponsor-Investigator, Emily de los Reyes, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005148
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: SLC6A1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AAV9.SLC6A1 Gene Therapy (Experimental)
  Interventions: Biological: AAV9.SLC6A1 Gene Therapy

INTERVENTIONS:
Biological: AAV9.SLC6A1 Gene Therapy — This is an open-label, single injection study of an AAV9 vector carrying the SLCA1 coding sequence delivered one time through an intrathecal injection.

SUMMARY:
This is gene therapy study of an AAV9 vector carrying the SLCA1 gene for SLC6A1 neurodevelopmental disorder.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of pathogenic mutation S295L in the SLC6A1 gene
* Ability to cooperate and complete assessments per determination of the physician and therapists

Exclusion Criteria:

* Serological evidence of HIV infection, or Hepatitis B or C infection
* Diagnosis of (or ongoing treatment) for an autoimmune disease
* Presence of a medical condition or extenuating circumstance that, in the opinion of the Sponsor-Investigator, might compromise the participant's ability to comply with the protocol required testing or procedures or compromise the participant's wellbeing, safety, or clinical interpretability
* Persistent leukopenia or leukocytosis (WBC ≤ 3.5 K/µL or ≥20.0 K/µL) or an absolute neutrophil count < 1.5K/µL
* Concomitant illness or requirement for chronic drug treatment that in the opinion of the Sponsor-Investigator creates unnecessary risks for gene transfer
* AAV9 binding antibody titers > 1:400 as determined by ELISA immunoassay
* Contraindications for intrathecal injection procedure (e.g. spina bifida, meningitis, or clotting abnormalities)
* Abnormal laboratory values in the clinically significant range upon normal values in the Nationwide Children's Hospital Laboratory. (GGT > 78 U/L, Bilirubin ≥ 3.0 mg/dL , Creatinine ≥ 1.8 mg/dL, Hgb < 8 or > 18 g/dL; WBC > 15,000 cells per mL)
* Family does not want to disclose participant's study participation with primary care physician and other medical providers.
* Bleeding disorder or any other medical conditions or circumstances in which intrathecal (IT) administration of the product or lumbar puncture (for collection of CSF) are contradicted according to local institutional policy
* Two consecutive aminotransaminase liver tests >3 times the upper limit of normal) at screening
* Contraindications for MRI scans (e.g., cardiac pacemaker, metal fragment or chip in the eye, aneurysm clip in the brain

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2028-08-25 (Estimated); Study Completion 2030-08-25 (Estimated)

PRIMARY OUTCOMES:
Monitoring for the development of unacceptable toxicity. | 3 years
  Unacceptable toxicity is defined as the occurrence of two or more unexpected Grade III or higher treatment-related toxicities that are at least possibly related to the product or procedure, as defined by CTCAE 5.0.

SECONDARY OUTCOMES:
Change the Autism Diagnostic Schedule (ADOS), Module 3, scores from baseline to 3 years following gene therapy. | 3 years
  Scores on the ADOS, Module 3, will be measured by a certified clinical evaluator.
Change the Vineland Adaptive Behaviour Scale (VABS) scores from baseline to 3 years following gene therapy. | 3 years
  Scores on the Vineland Adaptive Behaviour Scale (VABS) will be measured by a certified clinical evaluator.
Change the Child Behaviour Checklist scores from baseline to 3 years following gene therapy. | 3 years
  Scores on the Child Behaviour Checklist will be measured by a certified clinical evaluator.

CONTACTS AND LOCATIONS:
Overall Officials: Emily de los Reyes, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Due to this being an N = 1 study, providing IPD publicly would likely deidentify the participant.